CLINICAL TRIAL: NCT03311035
Title: LIFT Technique Versus Seton in Management of Anal Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanob Hosny, Resident doctor at General surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anal fistula
Record Dates: First submitted 2017-08-25; First posted 2017-10-16 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: Patients will be classified into two groups according to the surgical procedure performed as follows:
  * Group A: Patients undergoing cutting Seton.
  * Group B: Patients undergoing LIFT technique
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): patients undergoing ligation of intersphincteric fistula tract (LIFT technique)
  Interventions: Procedure: LIFT technique
- Group B (Experimental): patients undergoing Seton method
  Interventions: Procedure: Seton

INTERVENTIONS:
Procedure: Seton — The identification of the primary tract of the fistula and the placement of the thread can be performed in one single step. a non-absorbable, braided thread is inserted . After excision of the external opening and the extrasphincteric parts of the fistula, the thread is grasped and is pulled out of the anus .The thread is cut in two parts. The mucosa is incised over the muscular bridge . One thread is tied snugly around the muscle; the other is tied loosely .The snugly tied seton has to be replaced after 14 days to provide appropriate tension to cut slowly trough the muscle. This can easily be achieved with the second loosely tied seton . A new thread is folded in the middle and connected to the opened sling of the loose seton using a special knot shown in.The old thread is removed and in the same maneuver two new setons are placed. Again, one thread is tied snugly around the remaining portion of the sphincter muscle; the other is tied loosely .
  Arms: Group B
Procedure: LIFT technique — The internal opening was identified . The intersphincteric plane was entered via a curvilinear incision corresponding to the site of the internal opening at the intersphincteric groove. The intersphincteric plane was developed by meticulous scissor and diathermy dissection up to the tract. Once identified, a small, right-angled clamp was hooked underneath or a tape passed round it. the tract was then transfixed close to the internal sphincter with 2/0 polyglactin suture . Saline was gently injected through the external opening to confirm that the tract was no longer patent and it was then divided distal to the point of ligation . After light traction, a segment of the distal tract was excised and, if needed, any defect in the external sphincter was closed. The intersphincteric incision wound was re-approximated loosely with interrupted 2/0 Vicryl. Partial core-out of the fistula tract was performed from the external opening to the external sphincter.
  Arms: Group A

SUMMARY:
Abscesses and anal fistulas represent about 70% of perianal suppuration, with an estimated incidence of 1/10,000 inhabitants per year and representing 5% of queries in coloproctology.

Anal fistula is the chronic phase of anorectal infection is characterized by chronic purulent drainage or cyclic pain associated with acute relapse of the abscess followed by intermittent spontaneous decompression.

Perianal fistulas have a troublesome pathology. The most widely accepted theory is that anal abscess is caused by infection of an anal crypt gland. Suppuration moves from the anal gland to the inter-sphincteric space, forming an abscess leading to the development of a fistula. The incidence of fistula following an abscess is nearly 33%.

A fistula can cause pain, perianal swelling, discharge, bleeding, and other nonspecific symptoms.

The diagnosis of fistula-in-ano may include a digital rectal examination, endoanal ultrasound, fistulography, and MRI.

The management of the disease is difficult and sometimes a challenge for the surgeon.

The ideal treatment is based on three central principles: control of sepsis, closure of the fistula and maintenance of continence.

The management of complex fistulas needs to balance the outcomes of cure and continence. Success is usually determined by identification of the primary opening and dividing the least amount of muscle as possible.

There is a risk of sphincter muscle damage during fistulotomy, which can lead to an unacceptable risk of anal incontinence of varying degrees.

The surgical techniques described for the treatment of fistula-in-ano are fistulotomy, core-out fistulectomy, seton placement, endorectal advancement flap, injection of fibrin glue, insertion of a fistula plug, video-assisted anal fistula treatment (VAAFT) and ligation of the intersphincteric fistula tract (LIFT), Surgical techniques are composed of 2 broad categories, including sphincter sacrificing procedures, such as, fistulotomy, fistulectomy and cutting seton. and sphincter-preserving procedures, such as fibrin glue injection, fistula plug, rectal advancement flap, VAAFT and LIFT. In general, sphincter sacrificing procedures have high success rates but are associated with high rates of fecal incontinence. In contrast, sphincter-preserving procedures have more modest success rates but are associated with a relatively minimal risk of changes in continence.

While low transsphincteric fistulae are well-addressed by fistulotomy (i.e., lay-open technique) with minimal change in long-term bowel habits, fistulae which involve more than 30 % of the internal sphincter carry a substantial risk of fecal incontinence with this approach.

Endorectal advancement flap is technically difficult and associated with high recurrence rate up to 50% and risk of incontinence up to 35%.

Fibrin glue and anal fistula plug have a little effect on incontinence but are associated with high recurrence up to 60 % and are costive.

VAAFT is effective method but is highly costive.

Setons can be employed as cutting and non-cutting kinds as dividers or markers . A few types of setons used are the Ayurveda-medicated thread , braided sutures thread, rubber band , Penrose drains and cable tie seton . Seton material should be non-absorbable, from non-slippage material, comfortable and least irritant for the patient and equally ejective in causing focal reaction in the track, leading to fibrosis .

However, setons may cause patient discomfort, both from irritation and from persistent drainage. In addition the incontinence rate may reach 67%.

The ligation of intersphincteric fistula tract (LIFT) was first described by Rojanasakul and colleagues in 2007. Since then, this technique has become popular among providers due to its simple technical elements, particularly when compared to anorectal advancement flaps, and favorable success rate. Among the many studies published in the literature, the success rate after LIFT ranges from 40 to 95 %, with a recurrence rate of 6-28 % .3,5-28 In comparison, success after advancement flap ranges from 60 to 94 %.

DETAILED DESCRIPTION:
This study is a prospective study;

B) Methodology:

Patients will be classified into two groups according to the surgical procedure performed as follows:

* Group A: Patients undergoing cutting Seton.
* Group B: Patients undergoing LIFT technique.

Aim OF THE STUDY:

To compare between Seton and LIFT technique in management of anal fistula according to ;

1-Feasibility of the technique. 3-Postoperative pain and use of analgesia. 4-Healing time. 5-Recurrence rate. 6-Occurrence of fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will undergo LIFT technique and Seton for management of anal fistula at General surgery department - Assiut University

Exclusion Criteria:

* patients under age of 16 years old.
* patients with malignant fistula.
* patients with crohn's disease.
* patients with Tuberculosis.
* patients with intersphincteric fistula. Patients with anal fistula and anal incontinence

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-18 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of the fistula | Up to one year from last case
  re-appearance of pus discharge or pain after healing of the fistula

SECONDARY OUTCOMES:
Postoperative pain | up to 2 weeks postoperatively for each case
  intensity of postoperative pain according to the number of doses needed for analgesia
Fecal Incontinence | up to 2 months postoperatively for each case
  patient complaining of involuntary passage of flatus or stool and confirmed by Digital Rectal examination and Electromyography
Healing time of the wound | up to 3 months postoperatively for each case
  number of days needed for closure of skin at external opening

IPD SHARING:
Plan to Share IPD: Undecided
All patients were discharged with analgesics and stool softeners and received oral ofloxacin and metronidazole for 1 week. Before being discharged, the patients were shown how to clean their wound and were advised to take topical antibiotic ointment. After hospital discharge, patients were seen 2 week after the initial procedure. The second consultation was 2 weeks after the first visit and the third visit will be after 6 month from the operation and the fourth visit will be after one year from the operation .At each visit the patient was interviewed for clinical continence status. The intersphincteric incision wound was examined, the sites of the previous internal and external openings were palpated and sphincter tone was assessed. After healing, the patient was asked to return should any recurrent pain, swelling or discharge occur. All patients with a documented healed fistula were also contacted by telephone at the time of the present study to enquire of possible recurrence.

REFERENCES:
- [Background] Dudukgian H, Abcarian H. Why do we have so much trouble treating anal fistula? World J Gastroenterol. 2011 Jul 28;17(28):3292-6. doi: 10.3748/wjg.v17.i28.3292. PMID 21876616
- [Background] Xu Y, Tang W. Ligation of Intersphincteric Fistula Tract Is Suitable for Recurrent Anal Fistulas from Follow-Up of 16 Months. Biomed Res Int. 2017;2017:3152424. doi: 10.1155/2017/3152424. Epub 2017 Feb 8. PMID 28271064
- [Background] Chen HJ, Sun GD, Zhu P, Zhou ZL, Chen YG, Yang BL. Effective and long-term outcome following ligation of the intersphincteric fistula tract (LIFT) for transsphincteric fistula. Int J Colorectal Dis. 2017 Apr;32(4):583-585. doi: 10.1007/s00384-016-2723-2. Epub 2016 Nov 23. PMID 27878618
- [Background] Khadia M, Muduli IC, Das SK, Mallick SN, Bag L, Pati MR. Management of Fistula-In-Ano with Special Reference to Ligation of Intersphincteric Fistula Tract. Niger J Surg. 2016 Jan-Jun;22(1):1-4. doi: 10.4103/1117-6806.169818. PMID 27013849
- [Background] Mushaya C, Bartlett L, Schulze B, Ho YH. Ligation of intersphincteric fistula tract compared with advancement flap for complex anorectal fistulas requiring initial seton drainage. Am J Surg. 2012 Sep;204(3):283-9. doi: 10.1016/j.amjsurg.2011.10.025. Epub 2012 May 19. PMID 22609079
- [Background] Charua-Guindic L, Mendez-Moran MA, Avendano-Espinosa O, Jimenez-Bobadilla B, Charua-Levy E. [Complex anal fistula treated with cutting seton]. Cir Cir. 2007 Sep-Oct;75(5):351-6. Spanish. PMID 18158881
- [Background] Ye F, Tang C, Wang D, Zheng S. Early experience with the modificated approach of ligation of the intersphincteric fistula tract for high transsphincteric fistula. World J Surg. 2015 Apr;39(4):1059-65. doi: 10.1007/s00268-014-2888-1. PMID 25472892
- [Background] Zirak-Schmidt S, Perdawood SK. Management of anal fistula by ligation of the intersphincteric fistula tract - a systematic review. Dan Med J. 2014 Dec;61(12):A4977. PMID 25441733